CLINICAL TRIAL: NCT00240084
Title: Nesiritide and Vo2 Max in Heart Failure Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Scios, Inc. (Industry)
Responsible Party: Principal Investigator, Leway Chen, MD, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NES V02
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nesiritide infusion (Experimental): Single arm study. 24-hour infusion of B-type Natriuretic Peptide at a dose of 0.01 mcg/kg/minute.
  Interventions: Drug: nesiritide (Natrecor(TM))

INTERVENTIONS:
Drug: nesiritide (Natrecor(TM)) — administration of IV nesiritide

SUMMARY:
This research study, funded by Scios, Inc., and conducted by the Cardiology Division of the Department of Medicine at the University of Rochester School of Medicine and Dentistry investigates the potential benefit of nesiritide (brand name is Natrecor(TM))in improving exercise capacity in patients with heart failure (HF). Previous studies have shown beneficial hemodynamic and neurohumoral effects of nesiritide infusion in the therapy of decompensated heart failure. Other studies have demonstrated increases in endogenous BNP levels (normalized for exercise workload) in HF patients during and after exercise. However, trials involving the measurement of exercise capacity in this population following BNP administration are lacking. This is an experimental prospective, non-blinded, pilot study with a sample size of 20 patients, all serving as their own controls. This study involves off-label use of the drug nesiritide (indicated for IV treatment of NYHA Class II and III patients, and this study is enrolling Class II and III patients) and has received FDA approval, and an IND. Subjects are recruited from the population of referrals to the Strong Memorial Hospital Heart Failure and Transplantation clinical service, who meet all the inclusion criteria and none of the exclusion criteria may participate in the study. Enrolled study subjects perform an exercise VO2 max test, receive a 24 hour infusion of nesiritide and perform a second exercise VO2 max test.

DETAILED DESCRIPTION:
See above comments.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 with NYHA Class II or III heart failure
* Referred to Strong Memorial Hospital for consideration of heart transplant
* Male or female and infertile or using effective contraception with negative pregnancy test
* Capable of IV access
* Able to perform a maximal bicycle test and tolerate mouthpiece and nose clip
* Fully understands and has signed Informed Consent Form before study begins
* Endogenous BNP level of at least 100 pg/mL
* Current smokers smoking < 3 cigarettes / day. Smoking is not permitted within the hospital, ergo subjects would not be permitted to smoke during study participation.

Exclusion Criteria:

* NYHA Class i or IV heart failure
* Creatinine clearance < 30 ml/min, as determined within 2 weeks of the start of the study
* EF > 40%
* Evidence of primary lung disease
* Hypersensitivity to nesiritide or any of its' components
* Current smokers as defined by > 3 cigarettes / day
* Stroke within 3 months, myocardial infarction within 2 months, or any evidence of active myocardial ischemia
* Unwillingness ir inability to remain in the hospital overnight
* Clinical condition or laboratory abnormality which may increase risks associated with participation or interfere with result interpretation
* Any condition which would preclude heart transplantation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-07; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Peak VO2 | 24 hours
  The goal of this study is to determine whether a continuous 24-hour infusion of B-type Natriuretic Peptide at a dose of 0.01 mcg/kg/minute will produce a significant improvement in exercise capacity as defined by maximum oxygen consumption (VO2 peak).

CONTACTS AND LOCATIONS:
Overall Officials: Leway Chen, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States